CLINICAL TRIAL: NCT02316691
Title: B-cell Depletion Therapy With Rituximab for Thyroid Eye Disease
Acronym: BetTeRTED
Status: Terminated | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Niveditha Mohan, MD, Assistant Professor of Medicine, University of Pittsburgh
Other Study IDs: PRO14060524; UL1TR000005 (NIH)
Record Dates: First submitted 2014-12-08; First posted 2014-12-15 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Thyroid Eye Disease
Keywords: Graves Disease; Rituximab
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be used to determine longitudinal effect of B cell depletion on frequencies and functions of T helper subsets and memory B cells in blood. Any unused PBMC as well as serum obtained from these blood draws will be banked for future use in in vitro experiments.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thyroid Eye Disease: Blood samples will be drawn from subjects diagnosed with Thyroid Eye Disease. This study is observational. No interventions will be given as part of this study.

SUMMARY:
Thyroid eye disease (TED) is an autoimmune inflammation of the orbital tissues that develops in up to 50% of patients with Graves' disease. Although about 80% respond to IVGC initially, the relapse rate is high and about 75% require further surgery despite initial response. Although the natural history of TED is associated with spontaneous remissions after about 1 to 3 years, many irreversible serious ophthalmic and orbital complications can arise during this time. Therefore, there is a need for improved intervention strategies in the early active inflammatory phase of TED, to avoid progression to the cicatricial stage where disease manifestations can only be addressed in a rehabilitative fashion. The primary immunopathogenesis of Graves' disease is considered to be activation of B cells that then produce autoantibody against thyrotropin receptors in the thyroid (TRAb). Like in many autoimmune diseases, the inflammatory CD4+ T cell subset known as Th17 cells is also increased in blood of patients with active Graves' disease; the putative Th17 cytokine, IL-17, is also increased in serum and tears of TED patients. There is also an emerging pathogenic role for Th17 cells that co-express the chemokine receptor CXCR5 and drive autoantibody production. The contribution of Th17 cells to TED is not well defined. This study is an observational, longitudinal, prospective study of patients receiving treatment for thyroid eye disease.

DETAILED DESCRIPTION:
All enrolled subjects will receive Intravenous Glucocorticoid (IVGC) therapy, which is currently the standard of care for TED patients. Subjects will receive the IVGC therapy at a facility chosen by them and their physician. If their disease does not respond to IVGC therapy, they will receive rituximab and/or surgical decompression and/or radiation which is also currently standard of care at a facility chosen by them and their physician. Prior to initiation of treatment and during the course of treatment, study patients will get research labs done along with routine labs and fill out questionnaires regarding their disease symptoms.

We will obtain 30 mL or 2 tablespoons of blood from subjects at initial evaluation and approximately Wk4, Wk 12, Wk 26, Wk 38, and Wk 52 (this may vary depending on when the patient comes in for their follow up visits, but the schedule approximates what is typical for standard of care in these patients) for mechanistic studies.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent
2. Age 18 to 75 years of age
3. Diagnosis of Thyroid Eye Disease (TED) with a CAS of ≥ 3. (Thyroid status can be euthyroid, hyper or hypothyroid.)
4. Willingness to practice birth control for at least 12 months post treatment.
5. Normal organ function, except if abnormal due to tumor involvement.
6. Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.
7. Subject has provided written informed consent.
8. Documentation of CD20 + status (for B cell malignancies).
9. ANC: > 1000/mm3
10. Adequate bone marrow function as indicated by a total white blood cell count of > 4 x 109/, hemoglobin of > 7 g/dl or a platelet count >100,000/mm³
11. Adequate renal function as indicated by creatinine of <2.5.
12. Adequate liver function, as indicated by AST or ALT <2x Upper Limit of normal unless related to primary disease.

Exclusion Criteria:

Patients will be excluded from the study based on the following criteria:

1. Brittle insulin dependent diabetes [The term "brittle" refers to cases of diabetes in which there is an instability that leads to a disruption of life and often recurrent and/ or prolonged hospitalization]
2. Pregnant or nursing patients
3. Significant medical comorbidities that would make the risk of high dose steroids intolerable such as severe CHF, CAD, arrhythmias, renal insufficiency, infection or immune deficiency, systemic autoimmune disease, severe glaucoma etc.
4. Absolute neutrophil count < 1500/mm³.
5. Contraindication to use of rituximab
6. Positive PPD and/or Quantiferon Gold TB test without prior anti-tuberculous therapy; active TB
7. HIV or hepatitis infection or declined consent for HIV or hepatitis testing
8. Use of rituximab in the prior 24 months for any reason other than TED
9. Unwillingness to practice birth control for at least 12 months post treatment
10. Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment), or lactating.
11. Inability to comply with study and/or follow-up procedures.
12. History of HIV.
13. Presence of active infection.
14. Presence of CNS metastases.
15. New York Heart Association Classification III or IV heart disease (See Appendix D).
16. Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
17. History of psychiatric disorder.
18. At the Investigator's discretion, receipt of a live vaccine within 4 weeks prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be introduced during a clinic visit with one of the physicians who are investigators on this study. These will be subjects who are being referred for intravenous glucocorticoid (IVGC) therapy due to the severe nature of their thyroid eye disease.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-01; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Remission of disease activity (decrease in CAS of ≥ 2) at 26 weeks after first rituximab/placebo infusion | 26 weeks
  Remission of symptoms and disease activity by 26 weeks after the first dose of medication. Subjects will be followed for one year to assess relapse

SECONDARY OUTCOMES:
Remission of disease activity (decrease in CAS of ≥ 2) at 6 and 14 weeks after first rituximab/placebo infusion. | 6 weeks
  Remission of symptoms by week 6 after treatment and again at week 14.
Maintenance of CAS (defined as no worsening of CAS or requirement of other interventions such as surgical decompression/orbital radiation by 26 weeks after first rituximab/placebo infusion . | 26 weeks
  Maintaining an absence of symptoms and disease activity.
Improvement in disease activity, as measured by CAS as a continuous variable at 6, 14, 26, 38 and 52 weeks after first infusion of rituximab, | 1 year
  Improvement in symptoms and disease activity
ll adverse effects related to RTX | 1 year
  Tracking any adverse events or serious adverse events related to rituximab.

OTHER OUTCOMES:
Efficacy outcome as measured by Time to ≥ 2 points improvement on the CAS. | 1 year
  Time to ≥ 2 points improvement on the CAS.
Efficacy outcome as measured by Decrease in exophthalmos (measured in mm using the same Hertel exophthalmometer and same intercanthal distance for an individual patient). | 1 year
  Decrease in exophthalmos (measured in mm using the same Hertel exophthalmometer and same intercanthal distance for an individual patient).
Efficacy outcome | 1 year
  Decrease in lid aperture (distance between the lid margins in mm with patient looking in the primary position, sitting relaxed and with distant fixation).
Efficacy outcome as measured by Subjective diplopia score | 1 year
  Subjective diplopia score (0=no diplopia; 1=intermittent, i.e. diplopia in primary position of gaze, when tired or when first awakening; 2= inconstant, i.e. diplopia at extremes of gaze; 3=constant, i.e. continuous diplopia in primary or reading position).
Efficacy outcome as measured by Improvement in quality of life as measured by an SF-36 and GoQoL. | 1 year
  Improvement in quality of life as measured by an SF-36 and GoQoL.
Efficacy outcome as measured by Immunologic markers and mechanistic analyses to include studies of peripheral blood and thyroid B and T cells and autoantibody levels, thyroid volume, cellularity and function. | 1 year
  Immunologic markers and mechanistic analyses to include studies of peripheral blood and thyroid B and T cells and autoantibody levels, thyroid volume, cellularity and function.

CONTACTS AND LOCATIONS:
Overall Officials: Niveditha Mohan, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Bahn RS. Graves' ophthalmopathy. N Engl J Med. 2010 Feb 25;362(8):726-38. doi: 10.1056/NEJMra0905750. PMID 20181974
- [Result] Bartalena L, Baldeschi L, Dickinson A, Eckstein A, Kendall-Taylor P, Marcocci C, Mourits M, Perros P, Boboridis K, Boschi A, Curro N, Daumerie C, Kahaly GJ, Krassas GE, Lane CM, Lazarus JH, Marino M, Nardi M, Neoh C, Orgiazzi J, Pearce S, Pinchera A, Pitz S, Salvi M, Sivelli P, Stahl M, von Arx G, Wiersinga WM; European Group on Graves' Orbitopathy (EUGOGO). Consensus statement of the European Group on Graves' orbitopathy (EUGOGO) on management of GO. Eur J Endocrinol. 2008 Mar;158(3):273-85. doi: 10.1530/EJE-07-0666. No abstract available. PMID 18299459
- [Result] Yeatts RP. Quality of life in patients with Graves ophthalmopathy. Trans Am Ophthalmol Soc. 2005;103:368-411. PMID 17057811
- [Result] HALES IB, RUNDLE FF. Ocular changes in Graves' disease. A long-term follow-up study. Q J Med. 1960 Jan;29:113-26. No abstract available. PMID 14398978
- [Result] Stan MN, Garrity JA, Bahn RS. The evaluation and treatment of graves ophthalmopathy. Med Clin North Am. 2012 Mar;96(2):311-28. doi: 10.1016/j.mcna.2012.01.014. Epub 2012 Feb 22. PMID 22443978
- [Result] Wakelkamp IM, Bakker O, Baldeschi L, Wiersinga WM, Prummel MF. TSH-R expression and cytokine profile in orbital tissue of active vs. inactive Graves' ophthalmopathy patients. Clin Endocrinol (Oxf). 2003 Mar;58(3):280-7. doi: 10.1046/j.1365-2265.2003.01708.x. PMID 12608932
- [Result] Douglas RS, Gupta S. The pathophysiology of thyroid eye disease: implications for immunotherapy. Curr Opin Ophthalmol. 2011 Sep;22(5):385-90. doi: 10.1097/ICU.0b013e3283499446. PMID 21730841
- [Result] Tuscano JM, Harris GS, Tedder TF. B lymphocytes contribute to autoimmune disease pathogenesis: current trends and clinical implications. Autoimmun Rev. 2003 Mar;2(2):101-8. doi: 10.1016/s1568-9972(02)00148-9. PMID 12848966
- [Result] Shen S, Chan A, Sfikakis PP, Hsiu Ling AL, Detorakis ET, Boboridis KG, Mavrikakis I. B-cell targeted therapy with rituximab for thyroid eye disease: closer to the clinic. Surv Ophthalmol. 2013 May-Jun;58(3):252-65. doi: 10.1016/j.survophthal.2012.10.006. Epub 2012 Dec 17. PMID 23253433
- [Result] Gaffen SL. Recent advances in the IL-17 cytokine family. Curr Opin Immunol. 2011 Oct;23(5):613-9. doi: 10.1016/j.coi.2011.07.006. Epub 2011 Aug 16. PMID 21852080
- [Result] Peng D, Xu B, Wang Y, Guo H, Jiang Y. A high frequency of circulating th22 and th17 cells in patients with new onset graves' disease. PLoS One. 2013 Jul 11;8(7):e68446. doi: 10.1371/journal.pone.0068446. Print 2013. PMID 23874630
- [Result] Kim SE, Yoon JS, Kim KH, Lee SY. Increased serum interleukin-17 in Graves' ophthalmopathy. Graefes Arch Clin Exp Ophthalmol. 2012 Oct;250(10):1521-6. doi: 10.1007/s00417-012-2092-7. Epub 2012 Jul 1. PMID 22752189
- [Result] Huang D, Xu N, Song Y, Wang P, Yang H. Inflammatory cytokine profiles in the tears of thyroid-associated ophthalmopathy. Graefes Arch Clin Exp Ophthalmol. 2012 Apr;250(4):619-25. doi: 10.1007/s00417-011-1863-x. Epub 2011 Nov 30. PMID 22124787
- [Result] Ma CS, Deenick EK. Human T follicular helper (Tfh) cells and disease. Immunol Cell Biol. 2014 Jan;92(1):64-71. doi: 10.1038/icb.2013.55. Epub 2013 Oct 22. PMID 24145858
- [Result] Morita R, Schmitt N, Bentebibel SE, Ranganathan R, Bourdery L, Zurawski G, Foucat E, Dullaers M, Oh S, Sabzghabaei N, Lavecchio EM, Punaro M, Pascual V, Banchereau J, Ueno H. Human blood CXCR5(+)CD4(+) T cells are counterparts of T follicular cells and contain specific subsets that differentially support antibody secretion. Immunity. 2011 Jan 28;34(1):108-21. doi: 10.1016/j.immuni.2010.12.012. Epub 2011 Jan 6. PMID 21215658